CLINICAL TRIAL: NCT05952336
Title: Transmission of Respiratory Viruses in Households in The Gambia: a Longitudinal Cohort Study
Brief Title: Transmission of Respiratory Viruses in Households in The Gambia: a Longitudinal Cohort Study (TransVIR)
Acronym: TransVIR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical Research Council Unit, The Gambia (Other)
Collaborators: UK Research and Innovation (Other)
Responsible Party: Sponsor
Organization: London School of Hygiene and Tropical Medicine (Other)
Other Study IDs: SCC 22556
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Respiratory Viral Infection; SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary endpoints

* Incidence of symptomatic and asymptomatic infection with SARS-CoV-2 and other respiratory viruses as determined by molecular (e.g. PCR) and serological testing
* Associations between the magnitude and quality of mucosal and serum antibody responses to SARSCoV- 2 and protection from infection with SARS-CoV-2
* Associations between the magnitude and quality of T cell responses to SARS-CoV-2 and protection from infection with SARS-CoV-2 Secondary endpoints
* Secondary attack rate and household cumulative infection rate with SARS-CoV-2, influenza, RSV, and other respiratory viruses
* Seroincidence and seroprevalence of SARS-CoV-2 a determined by binding antibodies to SARS-CoV-2 spike and nucleocapsid
* Presence of risk factors for symptomatic and asymptomatic infection with respiratory viruses
* Antibody and T cell kinetics of SARS-CoV-2 following infection
* Associations between the magnitude and quality of antibody and T cell responses to seasonal coronaviruses and protection from infection with SARS-CoV-2
* Associations between infection with non-SARS-CoV-2 respiratory viruses and protection from infection with SARS-CoV-2
* Associations between upregulation of gene expression in the mucosa, including interferon stimulated genes (ISGs), and protection from infection with SARS-CoV-2

DETAILED DESCRIPTION:
A prospective, observational cohort study within households in West Coast Region and Kanifing Municipality, The Gambia. A total of 50 - 70 households will be recruited. All members of the household will be included other than those who do not meet the eligibility criteria or decline to consent for the study. Participants will be enrolled for a total of 52 weeks, undergoing weekly field visits, along with an enrolment visit (V1), 6-month visit (V2) and 12-month visit (V3), which will all be clinic based. Clinic visits will collect anthropometric, socio-demographic and clinical data (including risk for acquisition of SARS-CoV- 2). In addition, a combined throat and nose swab (TNS), nasal lining fluid (NLF) using a synthetic absorptive matrix (SAM) strip, and a blood sample will be taken. Weekly visits will be done at the participants' homes or work place. During these visits, TNS will be collected, along with the presence of symptoms consistent with respiratory viral infections. In addition, participants who have symptoms consistent with influenza-like-illnesses (ILI) will have unscheduled visits where clinical data and a TNS is collected, which will be tested in real time for SARS-CoV-2 using PCR. Participants will be informed of their results within 24 hours after this TNS sample is collected at unscheduled ILI visits. Positive results will be communicated to the Ministry of Health for their records and contact tracing. Weekly TNS from all household members of any positive SARS-CoV-2 case will also be tested in real time for SARS-CoV-2 for 4 weeks following the most recent SARS-CoV- 2 positive case in the household. All participants with symptomatic SARS-CoV-2 detected at an unscheduled ILI visit will be seen at an additional clinic visit (post-covid follow up), where further TNS, NLF and blood samples will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Households must:
* be located in Kanifing municipality or West coast region.
* have at least 5 consented members.
* include the household head as a consented participant.
* have household members that includes at least one adult and at least one child.

Participants must:

- provide informed consent/assent according to their age.

Exclusion Criteria:

-

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Households will be excluded from participation if they meet any of the following criteria:
  - have plans to move away from the study area within the following year.
  Participants will be excluded from participation if they meet any of the following criteria:
  * have plans to move away from study area within the following year.
  * active participant in another research study.
Sampling Method: Non-Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic and asymptomatic infection with SARS-CoV-2 and other respiratory viruses as determined by molecular (e.g. PCR) and serological testing | 12 months
  with SARS-Incidence of symptomatic and asymptomatic infection with SARS-CoV-2 and other respiratory viruses as determined by molecular (e.g. PCR) and serological testingCoV-2 and other respiratory viruses as determined by molecular (e.g. PCR) and serological testing
  * Associations between the magnitude and quality of mucosal and serum antibody responses to SARSCoV- 2 and protection from infection with SARS-CoV-2
  * Associations between the magnitude and quality of T cell responses to SARS-CoV-2 and protection from infection with SARS-CoV-2
Associations between the magnitude and quality of mucosal and serum antibody responses to SARSCoV- 2 and protection from infection with SARS-CoV-2 | 12 months
  Associations between the magnitude and quality of mucosal and serum antibody responses to SARSCoV- 2 and protection from infection with SARS-CoV-2
Associations between the magnitude and quality of T cell responses to SARS-CoV-2 and protection from infection with SARS-CoV-2 | 12 months
  Associations between the magnitude and quality of T cell responses to SARS-CoV-2 and protection from infection with SARS-CoV-2

SECONDARY OUTCOMES:
Secondary attack rate and household cumulative infection rate with SARS-CoV-2, influenza, RSV, and other respiratory viruses | 12 months
  Secondary attack rate and household cumulative infection rate with SARS-CoV-2, influenza, RSV, and other respiratory viruses infection rate with SARS-CoV-2, influenza, RSV, and other respiratory viruses
  * Seroincidence and seroprevalence of SARS-CoV-2 a determined by binding antibodies to SARS-CoV-2 spike and nucleocapsid
  * Presence of risk factors for symptomatic and asymptomatic infection with respiratory viruses
  * Antibody and T cell kinetics of SARS-CoV-2 following infection
  * Associations between the magnitude and quality of antibody and T cell responses to seasonal coronaviruses and protection from infection with SARS-CoV-2
  * Associations between infection with non-SARS-CoV-2 respiratory viruses and protection from infection with SARS-CoV-2
  * Associations between upregulation of gene expression in the mucosa, including interferon stimulated genes (ISGs), and protection from infection with SARS-CoV-2
Seroincidence and seroprevalence of SARS-CoV-2 a determined by binding antibodies to SARS-CoV-2 spike and nucleocapsid | 12 months
  Seroincidence and seroprevalence of SARS-CoV-2 a determined by binding antibodies to SARS-CoV-2 spike and nucleocapsid
Presence of risk factors for symptomatic and asymptomatic infection with respiratory viruses | 12 months
  Presence of risk factors for symptomatic and asymptomatic infection with respiratory viruses
Antibody and T cell kinetics of SARS-CoV-2 following infection | 12 months
  Antibody and T cell kinetics of SARS-CoV-2 following infection
Associations between the magnitude and quality of antibody and T cell responses to seasonal coronaviruses and protection from infection with SARS-CoV-2 | 12 months
  Associations between the magnitude and quality of antibody and T cell responses to seasonal coronaviruses and protection from infection with SARS-CoV-2
Associations between infection with non-SARS-CoV-2 respiratory viruses and protection from infection with SARS-CoV-2 | 12 months
  Associations between infection with non-SARS-CoV-2 respiratory viruses and protection from infection with SARS-CoV-2
Associations between upregulation of gene expression in the mucosa, including interferon stimulated genes (ISGs), and protection from infection with SARS-CoV-2 | 12 months
  Associations between upregulation of gene expression in the mucosa, including interferon stimulated genes (ISGs), and protection from infection with SARS-CoV-2

CONTACTS AND LOCATIONS:
Locations (1):
- Field study in the West Coast Region and Kanifing Municipality Clinical Services Department, MRCG MRC Unit The Gambia at LSHTM (Fajara) Laboratories at MRC Unit The Gambia at LSHTM (Fajara) Laboratories at The University of Sheffield, UK, Banjul, West Coast, The Gambia

IPD SHARING:
Plan to Share IPD: No